CLINICAL TRIAL: NCT01004744
Title: Feasibility of Pre-Surgical Intervention Studies for Evaluating Targeted Therapies for Breast Cancer
Brief Title: Pre-Surgical Intervention for Targeted Therapies for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Avon Foundation (Other)
Responsible Party: Principal Investigator, Katherine D. Crew, Assistant Professor of Medicine and Assistant Professor of Epidemiology, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAC0553
Record Dates: First submitted 2009-10-28; First posted 2009-10-30 (Estimated); Results first posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Invasive Breast Cancer
Keywords: Postmenopausal women; ER+; Estrogen positive; PR+; Progesterone positive
MeSH Terms: interventions — Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Presurgical oral anastrozole (Experimental): 1mg daily for two weeks in the interval between diagnostic breast biopsy and definitive breast surgery.
  Interventions: Drug: Anastrozole

INTERVENTIONS:
Drug: Anastrozole — 1mg PO daily for two weeks prior to scheduled surgery
  Other Names: Arimidex

SUMMARY:
The purpose of this study is to determine the feasibility of a short term administration of a targeted therapy (i.e., anastrozole) in women with newly diagnosed early invasive or non invasive breast cancer during the interval between their breast biopsy and surgery. Anastrozole is a form of hormonal therapy which is part of the standard treatment for hormone sensitive breast cancer in postmenopausal women. This clinical model is being used to evaluate the biologic effects of this drug on a specific molecular pathway called the PI3K/AKT signaling pathway.

DETAILED DESCRIPTION:
Several clinical models are being explored for use in the phase I/II evaluation of targeted therapies for breast cancer. Biological markers can be measured in early stage invasive cancers in a presurgical model involving a short term intervention. In this model, women with newly diagnosed early invasive breast cancer receive a study drug during the interval between diagnostic breast biopsy and surgical resection. Tumor tissue obtained from the biopsy and surgical specimens are used to measure pre and post treatment molecular markers, respectively. The main advantages of this model include the ability to obtain direct information on molecular response in tumor tissue and elucidate drug mechanisms of action, the large patient population to draw from with early stage breast cancer, and the lack of unnecessary invasive procedures.

We plan to conduct a pilot study of 10 postmenopausal women with newly diagnosed estrogen receptor (ER) positive invasive or non invasive breast cancer who will receive oral anastrozole 1mg daily for two weeks in the interval between diagnostic breast biopsy and definitive breast surgery. Patients will be identified by the breast surgeon or mammographer performing the breast biopsy. Patients with histologically confirmed ER+ invasive or non invasive breast cancer will be recruited by the medical oncologist and will start anastrozole two weeks prior to their scheduled surgery. The primary objective of this study is to demonstrate the feasibility of this presurgical model for evaluating targeted therapies for breast cancer. Secondary endpoints include changes in tissue levels of the proliferation marker Ki67 and proteins involved in PI3K/AKT signaling.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed operable ER+ and/or PR+ invasive breast cancer or ductal carcinoma in situ (DCIS), who undergo core needle biopsy followed by surgical excision at least 2 weeks after enrollment
* Postmenopausal status defined as cessation of menses for >1 year or FSH > 20 mIU/mL (within the past month)
* Age ≥ 21 years
* No prior chemotherapy, radiation therapy, or surgery within 6 months of study entry
* Signed informed consent

Exclusion Criteria:

* Treatment with other investigational drugs within 6 months of study entry
* Other serious intercurrent medical illness

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Crew, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients will be identified by the breast surgeon or mammographer performing the breast biopsy. Patients with histologically-confirmed ER+ invasive or non-invasive breast cancer will be recruited by the medical oncologist and will start anastrozole two weeks prior to their scheduled surgery.
Period: Overall Study
Arm/Group | Presurgical Oral Anastrozole
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Presurgical Oral Anastrozole
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 5
Age, Continuous [Median (Full Range); unit: years] | 66 [49 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects That Completed Oral Anastrozole 1mg Daily for Two Weeks in the Interval Between Diagnostic Breast Biopsy and Definitive Breast Surgery
Description: The number of subjects who complete oral anastrozole for the length of the study is analyzed. The subjects receive oral anastrozole 1mg daily for two weeks in the interval between the biopsy and the surgery.
Time Frame: Two weeks
Measure: Number; unit: participants
Arm/Group | Presurgical Oral Anastrozole
Number analyzed (Participants) | 10
participants | 10

ADVERSE EVENTS:
Arm/Group | Presurgical Oral Anastrozole
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Presurgical Oral Anastrozole (N=10)
Diarrhea (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 4
Hot flashes (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No